CLINICAL TRIAL: NCT00693407
Title: Activation of Endogenous Inhibitory Modulation During Gastric and Somatic Stimulation in Functional Dyspepsia Patients and Healthy Controls
Brief Title: Study of Endogenous Inhibitory Modulation During Gastric and Somatic Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: NMRC, Singapore (Unknown)
Responsible Party: Principal Investigator, Medicine, Medicine, National University Hospital, Singapore
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: D/07/088
Record Dates: First submitted 2008-06-05; First posted 2008-06-09 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Functional Dyspepsia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1, FD patients (Experimental): Eighty male and female FD patients according to Rome III criteria (Drossman, 2006), aged 18 to 70 years, will be recruited from primary and secondary care via advertisements and our referral networks
  Interventions: Procedure: gastric capsaicin with heterotopic stimulation/ distraction
- 2,Healthy controls (Experimental): Forty male and female healthy volunteers, aged 18 to 70 years without any gastrointestinal pathology or history of significant abdominal pain, bowel disorders, bloating or discomfort during the last 3 months will be recruited.
  Interventions: Procedure: gastric capsaicin with heterotopic stimulation/ distraction

INTERVENTIONS:
Procedure: gastric capsaicin with heterotopic stimulation/ distraction — The subjects are randomized to swallow either a capsaicin 0.50mg capsule or an identical placebo capsule with 100ml of water If after 15 minutes pain scores do not reach a minimum level of 30, a further double-blinded capsule of the same content will be swallowed with 100ml of water. This is repeated to a maximum of 8 capusles until pain with VAS >30 is reported.

SUMMARY:
Visceral hypersensitivity as evidence of central sensory sensitization is evident in many patients with functional disorders such as functional dyspepsia (FD) and irritable bowel syndrome (IBS). We recently demonstrated both somatic hypersensitivity and abnormal endogenous pain modulation in IBS, both of which indicate central sensitization as a crucial mechanism in IBS. Endogenous pain mechanisms regulate, fine-tune and integrate sensory and homeostatic, including neuroendocrine, immune, motor and autonomic nervous system processes. Hitherto, no studies have investigated the role endogenous pain modulation in FD. Abnormal modulation could explain several of the symptom complexes associated with FD and provide a rationale for exploration of new treatments.

The current study was designed to

1. investigate the gastric sensitivity in FD patients and healthy controls during gastric capsaicin stimulation
2. assess the endogenous pain inhibitory modulation system in FD patients and healthy controls during heterotopic stimulation

ELIGIBILITY:
Inclusion Criteria:

FD patients:

* Eighty male and female FD patients according to Rome III criteria (Drossman, 2006), aged 18 to 70 years, will be recruited from primary and secondary care via advertisements and our referral networks.
* FD discomfort or pain should be the most prominent symptom.
* Patients must have been off all FD and analgesic medication and any drugs potentially influencing sensory function for at least two weeks before study start and be able to remain off such medication for the duration of the study period.

Healthy controls:

* Forty male and female healthy volunteers, aged 18 to 70 years without any gastrointestinal pathology or history of significant abdominal pain, bowel disorders, bloating or discomfort during the last 3 months will be recruited.

Exclusion Criteria:

Exclusion criteria for both FD patients and healthy controls:

* Organic gastrointestinal or other significant systemic disease, including cardiovascular, dermatological, psychiatric, neurological and endocrine diseases. Patients with peptic ulcer scars are also excluded.
* Chronic or acute pain, except related to other functional syndromes (irritable bowel syndrome, chronic pelvic pain, fibromyalgia, migraine).
* H. pylori positive.
* Abdominal surgery, including gastric resection or cholecystectomy (except appendectomy)
* History of brain disease or brain surgery.
* Ongoing treatment with any drugs or need for drugs (or complementary medication) within last 14 days.
* Treatment with any investigational drug during the preceding 30 days.
* Ingestion of spicy, chilli pepper containing meal, or use of capsaicin skin cream in last 48 hours before start of study or any study day.
* Pregnancy or lactation.
* No written informed consent obtained from subject.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-09; Primary Completion 2011-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Differences between healthy controls and FD subjects in visceral pain scores. | within 2 hours of Capsaicin challenge

CONTACTS AND LOCATIONS:
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore, Singapore
  - National University of Singapore, Singapore, Singapore